CLINICAL TRIAL: NCT01748825
Title: A Phase I Study of Single-agent AZD1775 (MK-1775), a Wee1 Inhibitor, in Patients With Advanced Refractory Solid Tumors
Brief Title: AZD1775 for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naoko Takebe, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 130032; 13-C-0032
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-06

CONDITIONS: Solid Tumors
Keywords: AZD1775; Adavosertib; MK-1775; Refractory; Solid Tumors; Wee1 Inhibitor; Tyrosine Kinase
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- ARM 1 AZD1775 200 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 2 AZD1775 225 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 3 AZD1775 225 mg Twice Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 4 AZD1775 225 mg Twice Daily (week 1-only dosing) (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 5 AZD1775 250 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 6 AZD1775 300 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 7 AZD1775 300 mg Twice Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 8 AZD1775 400 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)
- ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily (Experimental)
  Interventions: Drug: MK-1775 (AZD1775)

INTERVENTIONS:
Drug: MK-1775 (AZD1775) — MK-1775 (AZD1775) is an inhibitor of Wee1-kinase.In preclinical models, MK-1775 selectively enhanced chemotherapy-induced death of cells deficient in tumor protein p53 (p53) signaling.
  Other Names: Adavosertib

SUMMARY:
BACKGROUND:

* Wee1 is a tyrosine kinase involved in the phosphorylation and inactivation of cyclin-dependent kinase 1 (CDK1/CDC2)-bound cyclin B, resulting in G2 cell cycle arrest in response to deoxyribonucleic acid (DNA) damage to allow time for DNA repair. Recent preclinical data additionally implicates Wee1 in maintenance of genomic integrity during S phase.
* Adavosertib (AZD1775) is a selective inhibitor of Wee1 kinase. Recent preclinical model data additionally show single agent anti-tumor activity in multiple cancer cell lines and tumor xenografts.
* Preliminary data show AZD1775 is tolerable at lower doses in combination with chemotherapeutic agents. We propose to demonstrate single-agent activity for AZD1775.

PRIMARY OBJECTIVE:

* To establish the safety and tolerability of single-agent AZD1775 in patients with refractory solid tumors
* To determine the pharmacokinetics of AZD1775 in patients with refractory solid tumors

SECONDARY OBJECTIVES:

* To determine the effect of AZD1775 on markers of DNA damage and apoptosis in tumor tissue and circulating tumor cells
* To evaluate the antitumor activity of AZD1775 in patients with refractory solid tumors

EXPLORATORY OBJECTIVES:

-To identify tumor genomic alterations and gene expression patterns potentially associated with AZD1775 antitumor activity

ELIGIBILITY:

* Patients must have histologically confirmed solid tumors for which all standard therapy known to prolong survival have failed, or for which standard therapies do not exist.
* No major surgery, radiation, or chemotherapy within 3 weeks or (5 half-lives, whichever is shorter) prior to entering the study.
* Adequate organ function

STUDY DESIGN:

* This study will follow a traditional 3+3 design.
* In Arm A starting at dose level 1, AZD1775 will be administered orally, twice a day (BID), for 5 doses (Day (D) 1-3) during each cycle. Starting at dose level 2 and onwards, AZD1775 will be administered orally, BID, for 5 doses for the first 2 weeks of each cycle (D1-3 and 8- 10). Each cycle is 21 days (+/- 1 day for scheduling).
* Once maximum tolerated dose (MTD) is established, 6 additional patients will be enrolled at the MTD to further evaluate that dose for pharmacokinetics (PK) and pharmacodynamics (PD) endpoints.
* A further expansion arm of 6 additional patients with documented tumors harboring breast cancer type 1 or 2 (BRCA)-1 or -2 mutations will also be enrolled at the MTD to further explore the safety of the agent and obtain preliminary evidence of activity in this patient population.
* Based on preliminary evidence of drug activity in an alternative once-daily dosing schedule, patients without a documented BRCA mutation will be accrued to a once-daily dosing schedule Arm B, with mandatory paired tumor biopsies at the maximum tolerated single daily dose, to further evaluate PD endpoints. AZD1775 will be administered orally once daily for 5 days (D1-5 and 8-12) during weeks 1 and 2 of each 21-day cycle (+/- 1 day for scheduling).
* During the escalation phase, tumor biopsies will be optional and will be evaluated for pharmacodynamic (PD) studies for evidence of Wee1 inhibition DNA damage and repair, and apoptosis (gamma H2A histone family member X (yH2AX), phosphorylated Nbs1 (pNbs1), Rad51, Rabbit polyclonal phospho-cyclin-dependent kinases (pTyr15-Cdk) and caspase 3). During the expansion phase, once MTD is reached, mandatory paired tumor biopsies will be pursued in up to 20 additional patients enrolled at the MTD to further evaluate PD endpoints.

DETAILED DESCRIPTION:
BACKGROUND:

* Wee1 is a tyrosine kinase involved in the phosphorylation and inactivation of cyclin-dependent kinase 1 (CDK1/CDC2)-bound cyclin B, resulting in G2 cell cycle arrest in response to deoxyribonucleic acid (DNA) damage to allow time for DNA repair. Recent preclinical data additionally implicates Wee1 in maintenance of genomic integrity during S phase.
* Adavosertib (AZD1775) is a selective inhibitor of Wee1 kinase. Recent preclinical model data additionally show single agent anti-tumor activity in multiple cancer cell lines and tumor xenografts.
* Preliminary data show AZD1775 is tolerable at lower doses in combination with chemotherapeutic agents. We propose to demonstrate single-agent activity for AZD1775.

PRIMARY OBJECTIVE:

* To establish the safety and tolerability of single-agent AZD1775 in patients with refractory solid tumors
* To determine the pharmacokinetics of AZD1775 in patients with refractory solid tumors

SECONDARY OBJECTIVES:

-To evaluate the antitumor activity of AZD1775 in patients with refractory solid tumors

EXPLORATORY OBJECTIVES:

-To determine the effect of AZD1775 on markers of DNA damage and apoptosis in tumor

tissue and circulating tumor cells

* To assess whether sufficient Wee1 inhibition is maintained throughout the therapeutic regimen
* To identify tumor genomic alterations and gene expression patterns potentially associated withAZD1775 antitumor activity

ELIGIBILITY:

* Patients must have histologically confirmed solid tumors for which all standard therapy known to prolong survival have failed, or for which standard therapies do not exist.
* No major surgery, radiation, or chemotherapy within 3 weeks or (5 half-lives, whichever is shorter) prior to entering the study.
* Adequate organ function

STUDY DESIGN:

* This study will follow a traditional 3+3 design.
* In Arm A starting at dose level 1, AZD1775 will be administered orally, twice a day (BID), for 5 doses (D1-3) during each cycle. Starting at dose level 2 and onwards, AZD1775 will be administered orally, BID, for 5 doses for the first 2 weeks of each cycle (D1-3 and 8- 10). Each cycle is 21 days (+/- 1 day for scheduling).
* Once maximum tolerated dose (MTD) is established, 6 additional patients will be enrolled at the MTD to further evaluate that dose for pharmacokinetics (PK) and pharmacodynamics (PD) endpoints.
* A further expansion arm of 6 additional patients with documented tumors harboring breast cancer type 1 or 2 (BRCA)-1 or -2 mutations will also be enrolled at the MTD to further explore the safety of the agent and obtain preliminary evidence of activity in this patient population.
* Based on preliminary evidence of drug activity in an alternative once-daily dosing schedule, patients without a documented BRCA mutation will be accrued to a once-daily dosing schedule Arm B, with mandatory paired tumor biopsies at the maximum tolerated single daily dose, to further evaluate PD endpoints. AZD1775 will be administered orally once daily for 5 days (D1-5 and 8-12) during weeks 1 and 2 of each 21-day cycle (+/- 1 day for scheduling).
* During the escalation phase, tumor biopsies will be optional and will be evaluated for pharmacodynamic (PD) studies for evidence of Wee1 inhibition DNA damage and repair, and apoptosis (gamma H2A histone family member X (yH2AX), phosphorylated Nbs1 (pNbs1), Rad51, Rabbit polyclonal phospho-cyclin-dependent kinases (pTyr15-Cdk) and caspase 3). During the expansion phase, once MTD is reached, mandatory paired tumor biopsies will be pursued in up to 20 additional patients enrolled at the MTD to further evaluate PD endpoints.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Patients must have histologically confirmed solid tumors for which all standard therapy known to prolong survival have failed or for which standard therapies do not exist.
* Patients must have measurable disease or evaluable disease for the escalation phase; for the 6 additional patients enrolled at maximum tolerated dose (MTD) for further evaluation of pharmacokinetics (PK) and pharmacodynamics (PD) endpoints (Expansion Cohort A). For the 6-patient breast cancer gene (BRCA)-mutation expansion cohort, patients must have measurable disease; however, tumor biopsies are optional. For Expansion Cohort B, patients must have tumor amenable to biopsy (excisional or incision biopsies of skin or head (H) & neck (N) lesions under visualization) and willingness to undergo a tumor biopsy or patient will be undergoing a procedure due to medical necessity during which the tissue may be collected, or tumor biopsy tissue from a previous research study or medical care is available for submission at registration. Criteria for the submission of tissue are:

  * Tissue must have been collected within 3 months prior to registration
  * Patient has not received any intervening therapy for their cancer since the collection of the tumor sample
  * Tumor tissue must meet the minimum requirements
* Patients must have completed any chemotherapy, radiation therapy, surgery, or biologic therapy greater than or equal to 3 weeks (or > 5 half-lives, whichever is shorter) prior to entering the study. Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in an exploratory Investigational New Drug (IND)/Phase 0 study or more than or equal to 1 week from palliative radiation therapy. Patients must have recovered to eligibility levels from prior toxicity or adverse events.
* Age greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky >60%)
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin >9 g/dL
  * total bilirubin less than or equal to 1.5 times institutional upper limit of normal
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) less than or equal to 3 times institutional upper limit of normal
  * creatinine less than or equal to 1.5 times institutional upper limit of normal OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
* The effects of Adavosertib (AZD1775) on the developing human fetus are unknown. For this reason and because molecular inhibitors of Wee1 kinase are known to be teratogenic, women of child-bearing potential (WoCBP) may be included only if acceptable contraception is in place for two weeks before study entry, for the duration of the treatment with the study drug, and for 2 months after the last dose of AZD1775. Male patients who are involved in the study must agree to avoid procreative and unprotected sex (i.e., by using acceptable forms of contraception) and must not donate sperm during the study and for 3 months after the last dose of AZD1775. Where the female partner is pregnant or not using effective birth control, men should be advised to abstain while in the study and for 3 months after the last dose of AZD1775. Female partners, who are of child-bearing potential, of men participating in clinical studies of AZD1775 will also be required to use effective contraceptive measures while their partner is on study drug and for 3 months thereafter. Male patients will be advised to arrange for the freezing of sperm samples prior to the start of the study should they wish to father children while on AZD1775 or during the 3 months after stopping AZD1775.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first of study drug and women should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
* Patients must be able to swallow whole tablets or capsules. Nasogastric or G-tube administration is not allowed. Any gastrointestinal disease which would impair ability to swallow, retain, or absorb drug is not allowed.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with prostate cancer can continue to receive treatment with gonadotropin-releasing hormone (GnRH) agonists while on study, as long as there is evidence of disease progression on therapy.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with known active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks following treatment of brain metastases are eligible to participate at the discretion of the principal investigator.
* Eligibility of subjects receiving any medications or substances with the potential to affect the activity or pharmacokinetics of AZD1775 will be determined following review by the principal investigator.
* Patients receiving any medications or substances that are inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4), or CYP3A4 substrates need to be reviewed by the principal investigator. Continuation of such medications will be at the discretion of the principal investigator. Concomitant use of aprepitant or fosaprepitant is prohibited. As grapefruit and Seville oranges are known to contain moderate inhibitors of CYP3A4, these fruits or their products (including marmalade, juice, etc.) should be avoided while taking AZD1775. The use of sensitive substrates of CYP3A4, such as atorvastatin, simvastatin and lovastatin, is also prohibited in this study. Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to: St. John's wort, kava, ephedra (mahung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of the study drugs on the developing fetus are unknown.
* Human immunodeficiency virus (HIV) positive patients on antiretroviral therapy are ineligible because of the potential for pharmacokinetics (PK) interactions.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoko Takebe, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe N, Broome M, Hunter T. Regulation of the human WEE1Hu CDK tyrosine 15-kinase during the cell cycle. EMBO J. 1995 May 1;14(9):1878-91. doi: 10.1002/j.1460-2075.1995.tb07180.x. PMID 7743995
- [Background] Dai Y, Grant S. New insights into checkpoint kinase 1 in the DNA damage response signaling network. Clin Cancer Res. 2010 Jan 15;16(2):376-83. doi: 10.1158/1078-0432.CCR-09-1029. Epub 2010 Jan 12. PMID 20068082
- [Background] Jazayeri A, Falck J, Lukas C, Bartek J, Smith GC, Lukas J, Jackson SP. ATM- and cell cycle-dependent regulation of ATR in response to DNA double-strand breaks. Nat Cell Biol. 2006 Jan;8(1):37-45. doi: 10.1038/ncb1337. Epub 2005 Dec 4. PMID 16327781
- [Derived] Do K, Wilsker D, Ji J, Zlott J, Freshwater T, Kinders RJ, Collins J, Chen AP, Doroshow JH, Kummar S. Phase I Study of Single-Agent AZD1775 (MK-1775), a Wee1 Kinase Inhibitor, in Patients With Refractory Solid Tumors. J Clin Oncol. 2015 Oct 20;33(30):3409-15. doi: 10.1200/JCO.2014.60.4009. Epub 2015 May 11. PMID 25964244
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0032.html

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM 1 AZD1775 200 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 200 mg by mouth (PO) once daily
- ARM 2 AZD1775 225 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 225 mg by mouth (PO) once daily
- ARM 3 AZD1775 225 mg Twice Daily: Cycle = 21 days. MK-1775 (AZD1775) 225 mg by mouth (PO) twice daily
- ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing): Cycle = 21 days. MK-1775 (AZD1775) 225 mg by mouth (PO) twice daily (week 1-only dosing)
- ARM 5 AZD1775 250 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 250 mg by mouth (PO) once daily
- ARM 6 AZD1775 300 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 300 mg by mouth (PO) once daily
- ARM 7 AZD1775 300 mg Twice Daily: Cycle = 21 days. MK-1775 (AZD1775) 300 mg by mouth (PO) twice daily
- ARM 8 AZD1775 400 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 400 mg by mouth (PO) once daily
- ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily: Cycle = 21 days. MK-1775 (AZD1775) 225mg by mouth (PO) twice daily
- ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily: Cycle = 21 days. MK-1775 (AZD1775) 300mg by mouth (PO) once daily
Period: Dose Escalation
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
Started | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 0 | 0
Completed | 4 | 2 | 6 | 2 | 2 | 4 | 2 | 3 | 0 | 0
Not Completed | 2 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Refused further treatment | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily | Total
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5 | 3 | 3 | 4 | 2 | 2 | 12 | 8 | 44
  >=65 years | 3 | 2 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.17 (19) | 58.13 (21.56) | 46.18 (19.26) | 48.4 (20.88) | 58.33 (4.1) | 56.97 (15.39) | 65.07 (10.51) | 63.13 (14.74) | 51.49 (10.82) | 65.59 (8.57) | 58 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 3 | 1 | 4 | 1 | 2 | 12 | 16 | 44
  Male | 3 | 3 | 5 | 0 | 2 | 2 | 2 | 1 | 1 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 12 | 19 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
  White | 3 | 3 | 5 | 2 | 3 | 5 | 3 | 3 | 12 | 15 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20 | 67
Tumor Type [Count of Participants; unit: Participants]
  Ovarian carcinoma | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4 | 6 | 14
  Endometrial carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Mesothelioma | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Breast carcinoma | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 2 | 8
  Alveolar soft part sarcoma | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Colon adenocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Leiomyosarcoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Pancreatic carcinoma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Prostate carcinoma | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Bladder carcinoma | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cervical carcinoma | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cholangiocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Endometrial carcinosarcoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Liposarcoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Pleomorphic sarcoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Synovial cell sarcoma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Uterine carcinosarcoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Non-small cell lung cancer | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Papillary serous ovarian carcinoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Squamous cell carcinoma | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Synovial cell carcinoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hepatocellular carcinoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Malignant fibrous histiocytoma sarcoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Salivary adenocarcinoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Ewing sarcoma | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Fallopian tube carcinoma | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sinonasal leiomyosarcoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Atypical granular cell paraspinal | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Peritoneal carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Embryonal cell | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Appendiceal carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Score (ECOG) [Count of Participants; unit: Participants] — ECOG: 0 is normal activity and 1 is symptoms, but ambulatory.
  Participants
    0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 7
    1 | 5 | 4 | 5 | 2 | 2 | 6 | 3 | 3 | 13 | 17 | 60
Median Number of Prior Therapies [Median (Full Range); unit: prior therapy] | 5 [2 to 13] | 3.5 [0 to 18] | 7.5 [1 to 9] | 11 [8 to 12] | 4 [4 to 4] | 3 [3 to 25] | 2 [2 to 4] | 15 [2 to 18] | 7 [2 to 18] | 8 [1 to 16] | 7 [0 to 25]

OUTCOME MEASURES:

1. Primary Outcome: To Establish the Safety and Tolerability of Single-agent AZD1775 in Patients With Refractory Solid Tumors
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx.19 mo/8 d for A1, 3 mo/28 d for A2, 10 mo/28 d for A3, 2 mo/14 d for A4, 20 mo/24 d for A5, 10 mo/23 d for A6, 4 mo/23 d for A7, 14 mo/11 d for A8, 15 mo/24 d for A9, and 77 mo/6 d for A10.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20
Participants | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20

2. Primary Outcome: Establish the Safety and Tolerability of Single-agent AZD1775 in Patients With Refractory Solid Tumors
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant but not immediately life-threatening. Grade 4 is life-threatening.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20
percentage of participants
  Grade 1-2 Anemia | 50 | 75 | 50 | 67 | 33 | 67 | 67 | 100 | 69 | 60
  Grade 3 Anemia | 33 | 25 | 17 | 67 | 0 | 33 | 33 | 67 | 15 | 30
  Grade 1-2 Lymphopenia | 50 | 75 | 67 | 67 | 33 | 67 | 67 | 67 | 54 | 80
  Grade 3 Lymphopenia | 50 | 25 | 17 | 33 | 33 | 17 | 33 | 67 | 8 | 25
  Grade 4 Lymphopenia | 0 | 0 | 0 | 33 | 0 | 0 | 33 | 0 | 0 | 10
  Grade 1-2 Neutropenia | 17 | 25 | 17 | 0 | 33 | 17 | 33 | 100 | 23 | 25
  Grade 3 Neutropenia | 17 | 25 | 0 | 0 | 0 | 0 | 33 | 67 | 8 | 30
  Grade 4 Neutropenia | 17 | 0 | 0 | 33 | 0 | 0 | 33 | 33 | 0 | 20

3. Primary Outcome: To Determine the Pharmacokinetics of AZD1775 in Patients With Refractory Solid Tumors.
Description: Mean plasma concentration (± standard deviation) of AZD1775 at baseline and after AZD1775 administration.
Time Frame: Pre-Treatment (Baseline) and Cycle 1 Days 1 and 3 (Arms 3 and 7) or Days 1 and 5 (Arms 1-2, 5-6, and 8)
Population: Participants are grouped by dose level. Arm 3 represents combined data for patients receiving 225 mg twice daily on days 1-2 and once on day 3 of each 21-day cycle and for patients receiving 225 mg twice daily on days 1-2 and 8-9 and once on days 3 and 10 (the latter includes both dose escalation and expansion phase patients); these data are combined because all of these patients received the same dose over the pharmacokinetic analysis period (cycle 1 days 1-3).
Measure: Mean (Standard Error); unit: nM
Groups:
- ARM 1 AZD1775 200 mg Once Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 200 mg once daily on cycle 1 days 1-5, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 2 AZD1775 225 mg Once Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 225 mg once daily on cycle 1 days 1-5, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 3 AZD1775 225 mg Twice Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 225 mg twice daily on cycle 1 days 1-2, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 5 AZD1775 250 mg Once Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 250 mg once daily on cycle 1 days 1-5, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 6 AZD1775 300 mg Once Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 300 mg once daily on cycle 1 days 1-5, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 7 AZD1775 300 mg Twice Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 300 mg twice daily on cycle 1 days 1-2, during which the plasma concentrations of AZD1775 were evaluated.
- ARM 8 AZD1775 400 mg Once Daily: Participants received AZD1775 (MK-1775; adavosertib) by mouth at a starting dose of 400 mg once daily on cycle 1 days 1-5, during which the plasma concentrations of AZD1775 were evaluated.
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily
Number analyzed (Participants) | 4 | 3 | 15 | 3 | 6 | 3 | 3
nM
  Pre-Treatment (Baseline) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 1, 1 hour post-dose | 135 (230) | 577 (248) | 262 (257) | 539 (236) | 426 (377) | 452 (402) | 641 (452)
  Cycle 1 Day 1, 2 hours post-dose | 402 (327) | 1017 (442) | 592 (354) | 766 (36) | 997 (703) | 878 (263) | 1407 (314)
  Cycle 1 Day 1, 4 hours post-dose | 600 (18) | 876 (420) | 661 (212) | 636 (43) | 979 (491) | 975 (361) | 1757 (351)
  Cycle 1 Day 1, 6 hours post-dose | 579 (152) | 677 (351) | 556 (210) | 462 (23) | 744 (412) | 780 (222) | 1537 (469)
  Cycle 1 Day 1, 8 hours post-dose | 416 (153) | 521 (232) | 422 (180) | 276 (101) | 604 (373) | 586 (209) | 1063 (256)
  Cycle 1 Day 3, pre-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 776 (341) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1560 (414) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 3, 1 hour post-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 983 (522) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2090 (403) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 3, 2 hours post-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1350 (673) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2440 (571) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 3, 4 hours post-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1440 (655) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2450 (583) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 3, 6 hours post-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1210 (633) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2190 (437) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 3, 8 hours post-dose | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1030 (509) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1980 (455) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775.
  Cycle 1 Day 5, pre-dose | 235 (55) | 325 (231) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 167 (48) | 237 (82) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 671 (156)
  Cycle 1 Day 5, 1 hour post-dose | 461 (108) | 961 (492) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 734 (88) | 774 (394) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1970 (301)
  Cycle 1 Day 5, 2 hours post-dose | 782 (83) | 1128 (465) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1135 (266) | 1697 (1062) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 3036 (572)
  Cycle 1 Day 5, 4 hours post-dose | 952 (66) | 1115 (440) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1114 (238) | 1638 (860) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2597 (211)
  Cycle 1 Day 5, 6 hours post-dose | 790 (95) | 985 (441) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 787 (177) | 1222 (491) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 2062 (511)
  Cycle 1 Day 5, 8 hours post-dose | 597 (79) | 892 (367) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 605 (147) | 965 (388) | NA (NA) — not applicable per protocol, as the protocol specified pharmacokinetic sample collection on days 1 and 3 for patients receiving twice-daily AZD1775 and on days 1 and 5 for patients receiving once-daily AZD1775. | 1697 (115)

4. Secondary Outcome: To Evaluate the Antitumor Activity of AZD1775 in Patients With Refractory Solid Tumors
Description: Objective Response is defined as a Complete Response + Partial Response and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 13 | 20
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4

5. Other Pre Specified Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: DLT is defined as an adverse event that is related (possibly, probably, or definitely) to administration of MK-1775 (Adavosertib (AZD1775). Examples are Grade ≥ 3 non-hematological toxicity, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with bleeding, Grade 3 fatigue of greater than 1 week duration, and failure to tolerate 100% of the dosing in the first cycle will be considered a DLT, etc.
Time Frame: First cycle (21 days) of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 3 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 19 mo. & 8 days for Arm 1, 3 mo. & 28 days for Arm 2, 10 mo. & 28 days for Arm 3, 2 mo. & 14 days for Arm 4, 20 mo. & 24 days for Arm 5, 10 mo. & 23 days for Arm 6, 4 mo. & 23 days for Arm 7, 14 mo. & 11 days for Arm 8, 15 mo. & 24 days for Arm 9, and 77 mo. & 6 days for Arm 10.
Groups:
- ARM 6 AZD1775 300 mg Once Daily; ARM 7 AZD1775 300 mg Twice Daily: Cycle = 21 days. MK-1775 (AZD1775) 300 mg by mouth (PO) twice daily
Arm/Group | ARM 1 AZD1775 200 mg Once Daily | ARM 2 AZD1775 225 mg Once Daily | ARM 3 AZD1775 225 mg Twice Daily | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) | ARM 5 AZD1775 250 mg Once Daily | ARM 6 AZD1775 300 mg Once Daily | ARM 7 AZD1775 300 mg Twice Daily | ARM 8 AZD1775 400 mg Once Daily | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/4 | 0/6 | 1/3 | 0/3 | 0/6 | 0/3 | 0/3 | 0/13 | 3/20
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/4 | 3/6 | 2/3 | 0/3 | 3/6 | 2/3 | 3/3 | 5/13 | 16/20
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 6/6 | 3/3 | 3/3 | 6/6 | 3/3 | 3/3 | 13/13 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 AZD1775 200 mg Once Daily (N=6) | ARM 2 AZD1775 225 mg Once Daily (N=4) | ARM 3 AZD1775 225 mg Twice Daily (N=6) | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) (N=3) | ARM 5 AZD1775 250 mg Once Daily (N=3) | ARM 6 AZD1775 300 mg Once Daily (N=6) | ARM 7 AZD1775 300 mg Twice Daily (N=3) | ARM 8 AZD1775 400 mg Once Daily (N=3) | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily (N=13) | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Gastrointestinal DIS;Hernia Wrapped around bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Disease Progression/Death
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive disease
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Neoplasms benign - Death
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Respiratory - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Surgical and medical procedures - Pleurodesis, pleurx (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Surgical and medical procedures - Thoracentesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 AZD1775 200 mg Once Daily (N=6) | ARM 2 AZD1775 225 mg Once Daily (N=4) | ARM 3 AZD1775 225 mg Twice Daily (N=6) | ARM 4 AZD1775 225 mg Twice Daily (Week 1-only Dosing) (N=3) | ARM 5 AZD1775 250 mg Once Daily (N=3) | ARM 6 AZD1775 300 mg Once Daily (N=6) | ARM 7 AZD1775 300 mg Twice Daily (N=3) | ARM 8 AZD1775 400 mg Once Daily (N=3) | ARM 9 Expansion Cohort 1: AZD1775 225 mg Twice Daily (N=13) | ARM 10 Expansion Cohort 2: AZD1775 300 mg Once Daily (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (9) | 4 (6)
Activated partial thromboplastin time prolonged (Investigations) | 3 (5) | 4 (5) | 1 (1) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 4 (7) | 0 (0) | 2 (6) | 3 (3) | 1 (1) | 1 (1) | 4 (6) | 3 (6)
Alkaline phosphatase increased (Investigations) | 4 (8) | 3 (3) | 3 (5) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 2 (4) | 4 (5) | 8 (13)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (7) | 3 (5) | 3 (5) | 3 (7) | 1 (1) | 4 (14) | 3 (5) | 3 (24) | 9 (23) | 17 (47)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 6 (14) | 11 (16)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (6) | 1 (1) | 4 (5) | 0 (0) | 1 (6) | 2 (3) | 1 (1) | 1 (2) | 3 (5) | 7 (9)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (8) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (6) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 7 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Creatinine increased (Investigations) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 2 (6) | 2 (3) | 2 (2) | 2 (3) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (5) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (13) | 2 (6) | 4 (21) | 2 (2) | 3 (11) | 4 (6) | 2 (2) | 3 (7) | 12 (47) | 14 (24)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 6 (7)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 5 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (8) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 13 (19)
Fever (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gastrointestinal disorders ? Other: Front teeth discomfort (unstable teeth, root canals involved)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 2 (11) | 1 (1) | 0 (0) | 1 (2) | 3 (4) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, Hepatobiliary disorders - fatty liver (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (5) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 2 (3) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 2 (2) | 0 (0) | 9 (21)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 6 (13) | 3 (6) | 2 (5) | 0 (0) | 2 (7) | 3 (4) | 5 (14) | 12 (36)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (14) | 2 (4) | 4 (6) | 2 (4) | 2 (4) | 4 (9) | 1 (1) | 3 (11) | 9 (14) | 15 (32)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (8) | 0 (0) | 1 (5) | 1 (1) | 3 (9) | 4 (4) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 2 (8) | 4 (8) | 5 (12)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5) | 2 (5) | 0 (0) | 1 (3) | 1 (2) | 3 (7) | 2 (2) | 2 (2) | 2 (3) | 8 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (8) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 3 (3) | 4 (6) | 6 (7)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Infections and infestations - MRSA at hospital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Investigations - Other, Gamma Glutamyl Transferase increased )GGT) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (12) | 3 (12) | 4 (9) | 3 (5) | 2 (10) | 4 (12) | 2 (3) | 2 (28) | 7 (11) | 18 (47)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Cramping of feet (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (12) | 4 (8) | 4 (17) | 2 (5) | 3 (11) | 2 (3) | 1 (1) | 3 (4) | 11 (49) | 16 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (peritoneal carcinomatosis)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Metastatic brain Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Burnt Smell/Smell sensitivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Nervous system disorder - "hangover" (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Nervous system disorders - "foggy and dazed" (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (7) | 1 (1) | 2 (3) | 3 (17) | 4 (11) | 7 (20)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 1 (1) | 3 (4) | 2 (4) | 1 (1) | 2 (10) | 2 (4) | 3 (23) | 6 (20) | 10 (31)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Renal and urinary disorders - prostatitis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cellulitis (R leg) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Skin and subcutaneous tissue disorders - port site red
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Surgical and medical procedure - tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, Atherosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (13) | 3 (6) | 5 (11) | 1 (3) | 2 (4) | 3 (3) | 1 (1) | 3 (3) | 9 (31) | 15 (25)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (2) | 3 (6) | 3 (6) | 1 (7) | 2 (3) | 3 (3) | 2 (23) | 7 (14) | 14 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT01748825/Prot_SAP_000.pdf
  • Informed Consent Form: Standard (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT01748825/ICF_001.pdf
  • Informed Consent Form: Genetic Analysis (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT01748825/ICF_002.pdf